CLINICAL TRIAL: NCT05747911
Title: Are Dietary Intake of Advanced Glycation End Products and Migraine Associated? A Case-control Study
Brief Title: Dietary Advanced Glycation End Products and Migraine
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Büşra Demirer, Ress. Asst., Karabuk University
Other Study IDs: Busra Demirer
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-02

CONDITIONS: Nutrition Disorders; Migraine Disorders
MeSH Terms: conditions — Nutrition Disorders; Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migraine
- Without Migraine

INTERVENTIONS:
Other:  — Groups will not be intervened. Only observational data will be used.

SUMMARY:
Is dietary intake of advanced glycation different between individuals with and without migraine? Is there a difference between the groups in terms of energy and nutrients? The answers to these questions are sought.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with episodic migraine by an experienced neurologist,
* For the control group, patients who were not diagnosed with migraine but applied to the headache outpatient clinic
* Volunteer

Exclusion Criteria:

* Being younger than 19 years and older than 64 years of age, having a history of cardiovascular disease, hypertension, diabetes, cancer, liver and kidney disease or other neurological disorder (epilepsy, multiple sclerosis, stroke, traumatic brain injury, etc.), secondary headache, antilipidemic and glucose taking intolerance medications or vitamin-mineral supplements, following a special diet, and consuming less than 800 kcal or more than 4000 kcal per day

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult individuals aged 19-64 who applied to Karabuk University Training and Research Hospital Neurology Clinic Headache Outpatient Clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Difference in dietary advanced glycation end products intake between groups | 2 months
  Is there a difference between the dietary intake of advanced glycation end products in individuals with migraine and healthy individuals? These values will be obtained from the food consumption records of the individuals. Intake of advanced glycation end product will be evaluated as ....kU/day.
  Is there a difference between the energy and nutrient intake of individuals with migraine and healthy individuals?

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No